CLINICAL TRIAL: NCT00869154
Title: Effect of Multidisciplinary Treatment in Patients With Mild Traumatic Brain Injury - a Randomized Controlled Trial
Brief Title: Multidisciplinary Treatment in Patients With Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSD 20425
Record Dates: First submitted 2009-02-24; First posted 2009-03-25 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Traumatic Brain Injury With Brief Loss of Consciousness
Keywords: Mild TBI; TBI (Traumatic Brain Injury); Traumatic Brain Injury; Injury, Brain, Traumatic; Injuries, Acute Brain; Brain Injuries, Traumatic; Acute Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Multidisciplinary outpatient rehabilitation with individual contacts and a psycho-educational group intervention at two outpatient rehabilitation clinics compared to follow-up by a general practitioner after a multidisciplinary examination.
Who Masked: Investigator
Masking Description: The baseline data were collected before randomization. The data collection at 12 months was conducted by postal self-report questionnaires, and for GOSE, an assistant who was blinded to the group allocation performed a telephone interview. Two independent persons, who were blinded for the groups and were unfamiliar with the aim and content of the study, entered the data into the SPSS database. A statistician, who did not participate in the treatment program and was blinded to the group allocation when the data were analyzed, controlled the data and performed the statistical analyses for RTW and the secondary outcomes.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary care follow up (Active Comparator): Multidisciplinary examination and follow up by the family doctor.
  Interventions: Behavioral: primary care follow up
- Multidisciplinary follow up (Experimental): Multidisciplinary examination and follow up by a multidisciplinary outpatient team.
  Interventions: Behavioral: Multidisciplinary follow up

INTERVENTIONS:
Behavioral: primary care follow up — Multidisciplinary examination, good advice from rehabilitation specialists and follow up by the family doctor.
  Other Names: Bergen Mild Traumatic Brain Injury Study.
  Arms: Primary care follow up
Behavioral: Multidisciplinary follow up — Multidisciplinary examination and follow up by rehabilitation specialists, a multidisciplinary team following an individual rehabilitation programs.
  Other Names: Bergen Mild Traumatic Brain Injury Study
  Arms: Multidisciplinary follow up

SUMMARY:
The aim of the study is to compare a multidisciplinary examination and follow up by rehabilitation program with a multidisciplinary examination, good advice and follow up by the family doctor.

Further on we will examine if there were differing clinical characteristics between patients who attended a planned follow-up session and those that failed to and Prognostic factors in mild traumatic brain injury patients after discharge from hospital.

DETAILED DESCRIPTION:
2 months after an acute mild traumatic brain injury (TBI) defined as Glasgow Coma Scale between 13 and 15. The patient will get a clinical examination by a specialist in rehabilitation medicine. Patient who wish or need a further follow up, are out of work or school, will be included and randomized to either a multidisciplinary follow up or primary care follow by their family doctor.

Both groups will got a multidisciplinary examination. The multidisciplinary team will work out a rehabilitation program and a report back to their family doctor.

Patient who got a multidisciplinary follow up will then get individual appointments and they will follow an educational program for 4 days. The topics are physical and psychical problems after TBI and problems in daily living and return to work. We will teach a way to accept and deal with their problems. A cognitive behavioural treatment or a psycho educative approach will be central in the treatment. The follow up period will be until 2 years if needed.

For booth groups we will make a registration of sick leave for 5 years. The Extended Glasgow Outcome Scale (GOS- E), Hospital Anxiety and Depression Scale (HAD), Rivermead post concussion symptoms questionnaire and Patient Global Impression of Change (PGIC) after 6 and 12 months.

Department of Economics at the University of Bergen will make cost-benefit analysis.

Further on we will examine if there were differing clinical characteristics between patients who attended a planned follow-up session and those that failed to, if sick leave or return to work could make a difference and Prognostic factors in mild traumatic brain injury patients after discharge from hospital. We also include demographic data, CT findings and clinical data based on information from the medical records, pain drawings and numeric rating scale for pain, Quality of Life and Subjective Health Complaints inventory. We got data about days on sick leave, diagnosis for sick leave and income for the first year before and after the injury from The Norwegian Labour and Welfare Service (NAV) through a third accredited agency Statistics Norway. From Statistics Norway we got additional information about education level and income.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted acute to Department of Neurosurgery ICD-10 diagnosed S06.0- S06.9
* Age 16 to 55 years
* Mild traumatic brain injury defined as Glasgow Coma Scale (GCS) between 13 and 15.

Exclusion Criteria:

* Earlier severe traumatic brain injury (GCS 8 or less).
* Serious psychiatric disease (ICD-10 diagnosed last two years).
* Known drug abuse (ICD-10 diagnosed last two years).
* Other serious illness which have a major impact of the outcome.
* Social client last two years as major income

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Return to work | 6 and 12 months after 1. multidisciplinary examination
  Sick leave for 5 years after injury

SECONDARY OUTCOMES:
GOSE | 6 and 12 months after 1. multidisciplinary examination
  Glasgow Outcome Scale Extended
Post-commotio symptoms (RPQ) | 12 months
  The Rivermead Post concussion symptoms Questionnaire
Patient's Global Impression of Change | 12 months
  Patient's Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sture Skouen, MD, PhD, Study Director — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Dept. physical medicine and rehabilitation, Bergen
  - Oslo University Hospital, Ullevål, Oslo

REFERENCES:
- See also: Publications from the project: Multidisciplinary outpatient treatment in patients with mild traumatic brain injury: A randomised controlled intervention study. — https://www.ncbi.nlm.nih.gov/pubmed/?term=vikane+e+not+diabetes